CLINICAL TRIAL: NCT02309528
Title: Chronic Kidney Disease Knowledge and Awareness Among American Indians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Stacey Jolly, Assistant Professor of Medicine; Staff Physician, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: K23DK091363 (NIH)
Record Dates: First submitted 2014-11-18; First posted 2014-12-05 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Educational computerized digital stories — computerized digital stories made by American Indians

SUMMARY:
Few educational intervention clinical trials have been conducted among those at risk for or with early chronic kidney disease. To the investigators' knowledge none have used digital storytelling as a means to deliver the educational message and have been conducted among American Indians, a group with high prevalence of chronic kidney disease and end stage kidney disease.

The aims of the research project are to:

1. Quantify levels of chronic kidney disease knowledge and awareness among American Indians.
2. Determine the effectiveness of a culturally tailored health presentation with computerized digital stories made by American Indians for improving chronic kidney disease knowledge and factors thought to be preventative of chronic kidney disease or its progression at baseline and follow-up in a pilot educational clinical intervention trial.

ELIGIBILITY:
Inclusion Criteria:

* Strong Heart Study or Strong Heart Family Study participant

Exclusion Criteria:

* End Stage Renal Disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Chronic Kidney Disease Knowledge | up to 12 months
  Survey of CKD Knowledge at baseline, post-intervention, 1-month follow up, 6 month follow up, and 12 month follow up

SECONDARY OUTCOMES:
Blood Pressure | Sept 2014-Sept 2015, baseline, 1-month, 6-month, and 12-month follow-up
  average resting blood pressure collected via automated BP machine which has 5 minute rest period, then collects BP at 1 minute intervals for 3 measurements, and then calculates an average
Self-reported doctor visits and hospitalizations | 1-month, 6-month, and 12-month follow-up
  Survey collection of self-reported doctor visits or hospitalizations
Self-reported new medical conditions | 1-month, 6-month, and 12-month follow-up
  Survey collection of self-reported new diagnoses (i.e. diabetes, hypertension)
Self-reported medication use and adherence | 1-month, 6-month, and 12-month follow-up
  Self-reported non-steroidal anti-inflammatory use and self-reported medication adherence of diabetes and/or blood pressure medications via the Morisky Medication Adherence Scale (MMAS-4)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States